CLINICAL TRIAL: NCT07110779
Title: Telenursing in Coronary Artery Disease: Randomized Clinical Trial and Patient Collaboration
Brief Title: Telenursing in Coronary Artery Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fernanda Maria Alves Lima (Other)
Collaborators: Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other)
Responsible Party: Sponsor-Investigator, Fernanda Maria Alves Lima, Collaborating professor, UPECLIN HC FM Botucatu Unesp
Organization: UPECLIN HC FM Botucatu Unesp (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TELENURS_CAD
Record Dates: First submitted 2025-07-21; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases
Keywords: coronary artery disease; cardiovascular diseases; telenursing; digital health; nursing
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telenursing consultation (Experimental): The intervention consists of telenursing appointments held at three points in time: one, three and five months after the first appointment.
  Interventions: Behavioral: Telenursing consultation
- Traditional follow-up (No Intervention): A final face-to-face evaluation will be conducted six months after the angioplasty to assess adherence to treatment and understanding of the coronary artery disease.

INTERVENTIONS:
Behavioral: Telenursing consultation — Telenursing consultations, which will be carried out via telephone calls, video calls, or messaging platforms, will be held between one, three, and five months after the first consultation. The North American Nursing Diagnosis Association (NANDA-I), the Nursing Outcomes Classification (NOC), and the Nursing Interventions Classification (NIC) taxonomies will be used to structure these consultations.
  Arms: Telenursing consultation

SUMMARY:
The aim of this research is to determine whether follow-up through telehealth consultations can enhance adherence to medication and increase knowledge about heart disease in patients with coronary artery disease (CAD) who have undergone coronary angioplasty. It can include individuals of any sex or gender, aged over 18, and with access to communication devices such as a cell phone, tablet, or internet-enabled computer. The main questions to be answered are:

* Does follow-up of patients with CAD through telenursing consultations improve adherence to the proposed treatment?
* Does the follow-up of patients with CAD, through telenursing consultations, improve knowledge about heart disease? The researchers will compare these patients with others who will be followed up as usual at the hospital to determine which group shows better adherence to drug treatment and greater knowledge about heart disease. The participants will have telenursing consultations at three intervals: one, three, and five months after the initial consultation. After six months from the first interview, both groups will be assessed. They will also be invited to participate in an activity to share their experiences and identify research priorities in the field, with the option to collaborate on future research.

DETAILED DESCRIPTION:
In the face of the global digital transformation, the leadership role of nurses is essential for developing digital health skills and implementing innovative strategies. In the context of coronary artery disease (CAD), telenursing has emerged as a crucial care strategy for monitoring patients, managing risk factors, promoting self-care, and enhancing quality of life.

The researchers will examine the prevalence of comorbidities and risk factors for cardiovascular disease (CVD) in the two study groups. They will also compare adherence to the proposed treatment and knowledge about CAD. Finally, they will draw up a protocol for telenursing consultations for patients with CAD undergoing coronary angioplasty. This protocol will be used at the institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angioplasty who have access to communication devices (mobile phone, tablet or computer with internet access).

Exclusion Criteria:

* Patients with serious comorbidities that prevent remote monitoring, those without access to the necessary technology for remote nursing, and those with a diagnosis that prevents communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
CADE-Q SV score | From the first appointment after coronary angioplasty until six months afterwards.
  The knowledge score regarding coronary artery disease (CAD) will be calculated using the Coronary Artery Disease Education Questionnaire Short Version (CADE-Q SV). This consists of 20 questions divided into five categories: clinical condition, risk factors, exercise, nutrition, and psychosocial risk. One point is awarded for each correct answer, with a maximum score of 20 points. The questionnaire aims to identify areas of low knowledge.
MTA score | From the first appointment after coronary angioplasty until six months afterwards.
  Adherence to the proposed treatment will be calculated using the Measure of Treatment Adherence (MTA) instrument. This consists of seven questions, with answers obtained using a six-point Likert scale. Adherence to treatment is determined by adding the values of each answer and dividing by the total number of items. Patients with an arithmetic mean score between one and four are considered non-adherent. Those with a score between five and six are considered adherent.

SECONDARY OUTCOMES:
Blood pressure | At the first consultation after coronary angioplasty, and six months later.
  Blood pressure measured in millimeters of mercury
Heart rate | At the first consultation after coronary angioplasty, and six months later
  Heart rate measured in beats per minute
Respiratory rate | At the first consultation after coronary angioplasty, and six months later
  Respiratory rate measured in movements per minute
Temperature | At the first consultation after coronary angioplasty, and six months later
  Temperature measured in degrees Celsius
Capillary blood glucose | At the first consultation after coronary angioplasty, and six months later
  Capillary blood glucose measured in milligrams per deciliter
Weight | At the first consultation after coronary angioplasty, and six months later
  Weight measured in kilograms
Height | At the first consultation after coronary angioplasty, and six months later
  Height measured in meters
Body Mass Index | At the first consultation after coronary angioplasty, and six months later
  Body mass index measured in kilograms per square meter
Waist | At the first consultation after coronary angioplasty, and six months later
  Waist circumference measured in centimeters
Hip | At the first consultation after coronary angioplasty, and six months later
  Hip circumference measured in centimeters
Waist-to-Hip Ratio | At the first consultation after coronary angioplasty, and six months later
  Waist-to-hip ratio calculated by dividing waist measurement by hip measurement

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda MA Lima, PhD, Principal Investigator — Universidade Estadual Paulista "Júlio de Mesquita Filho" - Unesp
Locations (1):
- Faculdade de Medicina de Botucatu - UNESP, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be preserved in accordance with the institution's repository policy and will be made available in the open access repository itself and presented at scientific conferences in the field, as well as publications in journals, keeping sensitive data anonymous.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: August 2025 - October 2026
Access Criteria: Access to research data by external parties will only be authorized upon prior request to the project's managing researcher. Data linked to manuscripts submitted or in the process of being submitted will be shared after acceptance and publication.

REFERENCES:
- [Background] Borba LO, Capistrano FC, Ferreira ACZ, Kalinke LP, Mantovani MF, Maftum MA. Adaptation and validation of the Measuring of Treatment Adherence for mental health. Rev Bras Enferm. 2018;71(suppl 5):2243-2250. doi: 10.1590/0034-7167-2017-0796. English, Portuguese. PMID 30365790
- [Background] Delgado AB, Lima ML. Contributo para a validação concorrente de uma medida de adesão aos tratamentos. Psicol Saúde Doenças. 2001; 2(2):81-100. Available from: https://scielo.pt/pdf/psd/v2n2/v2n2a06.pdf
- [Background] Ghisi GL, Durieux A, Manfroi WC, Herdy AH, Carvalho Td, Andrade A, Benetti M. Construction and validation of the CADE-Q for patient education in cardiac rehabilitation programs. Arq Bras Cardiol. 2010 Jun;94(6):813-22. doi: 10.1590/s0066-782x2010005000045. Epub 2010 May 7. English, Portuguese. PMID 20464275
- [Background] Ghisi GLM, Chaves GSS, Loures JB, Bonfim GM, Britto R. Validation of the Brazilian-Portuguese Version of a Short Questionnaire to Assess Knowledge in Cardiovascular Disease Patients (CADE-Q SV). Arq Bras Cardiol. 2018 Dec;111(6):841-849. doi: 10.5935/abc.20180169. Epub 2018 Sep 21. PMID 30281691
- [Background] Nygaard A, Halvorsrud L, Linnerud S, Grov EK, Bergland A. The James Lind Alliance process approach: scoping review. BMJ Open. 2019 Aug 30;9(8):e027473. doi: 10.1136/bmjopen-2018-027473. PMID 31473612
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Pereira SM, Barreto ML. Estudos de intervenção. In: Filho NA, Barreto ML. Epidemiologia & Saúde: Fundamentos, Métodos, Aplicações. 1ª ed. Rio de Janeiro: Guanabara Koogan; 2012. p. 215-24.
- [Background] Bensenor IM, Goulart AC, Thomas GN, Lip GYH; NIHR Global Health Research Group on Atrial Fibrillation Management. Patient and Public Involvement and Engagement (PPIE): first steps in the process of the engagement in research projects in Brazil. Braz J Med Biol Res. 2022 Jul 25;55:e12369. doi: 10.1590/1414-431X2022e12369. eCollection 2022. PMID 35894383
- [Background] Oliver K, Kothari A, Mays N. The dark side of coproduction: do the costs outweigh the benefits for health research? Health Res Policy Syst. 2019 Mar 28;17(1):33. doi: 10.1186/s12961-019-0432-3. PMID 30922339
- [Background] Brett J, Staniszewska S, Mockford C, Herron-Marx S, Hughes J, Tysall C, Suleman R. A systematic review of the impact of patient and public involvement on service users, researchers and communities. Patient. 2014;7(4):387-95. doi: 10.1007/s40271-014-0065-0. PMID 25034612
- [Background] Modigh A, Sampaio F, Moberg L, Fredriksson M. The impact of patient and public involvement in health research versus healthcare: A scoping review of reviews. Health Policy. 2021 Sep;125(9):1208-1221. doi: 10.1016/j.healthpol.2021.07.008. Epub 2021 Jul 24. PMID 34376328
- [Background] Russell J, Fudge N, Greenhalgh T. The impact of public involvement in health research: what are we measuring? Why are we measuring it? Should we stop measuring it? Res Involv Engagem. 2020 Oct 27;6:63. doi: 10.1186/s40900-020-00239-w. eCollection 2020. PMID 33133636
- [Background] Gibson A, Britten N, Lynch J. Theoretical directions for an emancipatory concept of patient and public involvement. Health (London). 2012 Sep;16(5):531-47. doi: 10.1177/1363459312438563. Epub 2012 Apr 25. PMID 22535648
- [Background] Hughes M, Duffy C. Public involvement in health and social sciences research: A concept analysis. Health Expect. 2018 Dec;21(6):1183-1190. doi: 10.1111/hex.12825. Epub 2018 Aug 29. PMID 30159960
- [Background] Ocloo J, Garfield S, Franklin BD, Dawson S. Exploring the theory, barriers and enablers for patient and public involvement across health, social care and patient safety: a systematic review of reviews. Health Res Policy Syst. 2021 Jan 20;19(1):8. doi: 10.1186/s12961-020-00644-3. PMID 33472647
- [Background] Padilha JC, Santos VB, Lopes CT, Lopes JL. Prevalence of pharmacological adherence in patients with coronary artery disease and associated factors. Rev Lat Am Enfermagem. 2021 Sep 3;29:e3464. doi: 10.1590/1518-8345.4554.3464. eCollection 2021. PMID 34495187
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] Saki M, Najmi S, Gholami M, Ebrahimzadeh F, Pour FJ. The effect of patient-centered education in adherence to the treatment regimen in patients with coronary artery disease. J Vasc Nurs. 2022 Mar;40(1):28-34. doi: 10.1016/j.jvn.2021.10.003. Epub 2021 Oct 27. PMID 35287831
- [Background] Sefidi N, Assarroudi A, Zandi Z, Malkemes SJ, Rakhshani MH, Abbaszade A, Sahebkar M. Evaluating the effects of telenursing on patients' activities of daily living and instrumental activities of daily living after myocardial infarction: A randomized controlled trial study. Geriatr Gerontol Int. 2022 Aug;22(8):616-622. doi: 10.1111/ggi.14426. Epub 2022 Jun 22. PMID 35734811
- [Background] Cunha DCPTD, Rossi LA, Dessote CAM, Bolela F, Dantas RAS. Evolution of self-care in patients with heart failure at the first outpatient return and three months after hospital discharge. Rev Lat Am Enfermagem. 2021 Jul 19;29:e3440. doi: 10.1590/1518-8345.4364.3440. eCollection 2021. PMID 34287539
- [Background] Nava LF, Duarte TTP, Lima WL, Magro MCS. Monitoramento avançado de enfermagem: pacientes de risco na atenção primária. Esc Anna Nery 2022; 26: e20210282. DOI: https://doi.org/10.1590/2177-9465-EAN-2021-0282
- [Background] Abraham C, Jensen C, Rossiter L, Dittman Hale D. Telenursing and Remote Patient Monitoring in Cardiovascular Health. Telemed J E Health. 2024 Mar;30(3):771-779. doi: 10.1089/tmj.2023.0187. Epub 2023 Sep 8. PMID 37682280
- [Background] Nurmeksela A, Pihlainen V, Kettunen T, Laukkanen J, Peltokoski J. Nurse-led counseling for coronary artery disease patients: A 1-year follow-up study. Nurs Health Sci. 2021 Sep;23(3):678-687. doi: 10.1111/nhs.12852. Epub 2021 Jun 3. PMID 33991019
- [Background] Sousa VLP, Dourado Junior FW, Anjos SJSBD, Moreira ACA. Nursing teleconsultation in primary health care: scoping review. Rev Lat Am Enfermagem. 2024 Sep 2;32:e4329. doi: 10.1590/1518-8345.7212.4329. eCollection 2024. PMID 39230178
- [Background] Iyamu I, Xu AXT, Gomez-Ramirez O, Ablona A, Chang HJ, Mckee G, Gilbert M. Defining Digital Public Health and the Role of Digitization, Digitalization, and Digital Transformation: Scoping Review. JMIR Public Health Surveill. 2021 Nov 26;7(11):e30399. doi: 10.2196/30399. PMID 34842555
- [Background] Fatehi F, Samadbeik M, Kazemi A. What is Digital Health? Review of Definitions. Stud Health Technol Inform. 2020 Nov 23;275:67-71. doi: 10.3233/SHTI200696. PMID 33227742
- [Background] Lapão LV. A Enfermagem do Futuro: combinando Saúde Digital e a Liderança do Enfermeiro. Rev. Latino-Am. Enfermagem. 2020; 28:e3338. DOI: http://dx.doi.org/10.1590/1518-8345.0000-3338
- [Background] Sousa SM, Bernardino E, Peres AM, Martins MM, Goncalves LS, Lacerda MR. The role of nurses in the integration of care for people with chronic noncommunicable diseases. Rev Esc Enferm USP. 2021 Sep 6;55:e20200131. doi: 10.1590/1980-220X-REEUSP-2020-0131. eCollection 2021. English, Portuguese. PMID 34495207
- [Background] Marcon SS, Ganassin GS, Arruda GO, Téston EF, Barreto MS, Marquete VF, Ferreira PC. Intervenção educativa no local de trabalho: promoção da saúde e prevenção cardiovascular com homens metalúrgicos. Rev. Baiana Enferm. 2021; 35: e 38619. DOI: https://doi.org/10.18471/rbe.v35.38619
- [Background] Arruda GO, Marcon SS, Peruzzo HE, Ruiz AGB, Back IR, Nass EMA, et al. Intervenção educativa em homens com diabetes mellitus: efeitos sobre comportamentos e perfil antropométrico. Acta Paul Enferm. 2020; 33: eAPE20190128. DOI: https://doi.org/10.37689/acta-ape/2020AO0128
- [Background] Arruda JA, Lemke VG, Mariani Jr. J, Barbosa AHP, Quadros AS, Pedra C et al. Posicionamento da Sociedade Brasileira de Cardiologia e da Sociedade Brasileira de Hemodinâmica e Cardiologia Intervencionista sobre Centro de Treinamento e Certificação Profissional em Hemodinâmica e Cardiologia Intervencionista - 2020. Arq Bras Cardiol. 2020; 114(1):137-93. DOI: https://doi.org/10.36660/abc.2019084
- [Background] Correction to: 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e649-e650. doi: 10.1161/CIR.0000000000000725. Epub 2019 Sep 9. No abstract available. PMID 31498691
- [Background] O'Donnell MJ, Chin SL, Rangarajan S, Xavier D, Liu L, Zhang H, Rao-Melacini P, Zhang X, Pais P, Agapay S, Lopez-Jaramillo P, Damasceno A, Langhorne P, McQueen MJ, Rosengren A, Dehghan M, Hankey GJ, Dans AL, Elsayed A, Avezum A, Mondo C, Diener HC, Ryglewicz D, Czlonkowska A, Pogosova N, Weimar C, Iqbal R, Diaz R, Yusoff K, Yusufali A, Oguz A, Wang X, Penaherrera E, Lanas F, Ogah OS, Ogunniyi A, Iversen HK, Malaga G, Rumboldt Z, Oveisgharan S, Al Hussain F, Magazi D, Nilanont Y, Ferguson J, Pare G, Yusuf S; INTERSTROKE investigators. Global and regional effects of potentially modifiable risk factors associated with acute stroke in 32 countries (INTERSTROKE): a case-control study. Lancet. 2016 Aug 20;388(10046):761-75. doi: 10.1016/S0140-6736(16)30506-2. Epub 2016 Jul 16. PMID 27431356
- [Background] Lanas F, Avezum A, Bautista LE, Diaz R, Luna M, Islam S, Yusuf S; INTERHEART Investigators in Latin America. Risk factors for acute myocardial infarction in Latin America: the INTERHEART Latin American study. Circulation. 2007 Mar 6;115(9):1067-74. doi: 10.1161/CIRCULATIONAHA.106.633552. PMID 17339564
- [Background] Teo KK, Rafiq T. Cardiovascular Risk Factors and Prevention: A Perspective From Developing Countries. Can J Cardiol. 2021 May;37(5):733-743. doi: 10.1016/j.cjca.2021.02.009. Epub 2021 Feb 19. PMID 33610690
- [Background] Feliciano SCDC, Villela PB, Oliveira GMM. Association between Mortality from Chronic Noncommunicable Diseases and Human Development Index in Brazil between 1980 and 2019. Arq Bras Cardiol. 2023 Apr 21;120(4):e20211009. doi: 10.36660/abc.20211009. eCollection 2023. English, Portuguese. PMID 37098983
- [Background] Mansur AP, Favarato D. Cardiovascular and Cancer Death Rates in the Brazilian Population Aged 35 to 74 Years, 1996-2017. Arq Bras Cardiol. 2021 Aug;117(2):329-340. doi: 10.36660/abc.20200233. English, Portuguese. PMID 34495229
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Anderson CAM, Arora P, Avery CL, Baker-Smith CM, Beaton AZ, Boehme AK, Buxton AE, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Fugar S, Generoso G, Heard DG, Hiremath S, Ho JE, Kalani R, Kazi DS, Ko D, Levine DA, Liu J, Ma J, Magnani JW, Michos ED, Mussolino ME, Navaneethan SD, Parikh NI, Poudel R, Rezk-Hanna M, Roth GA, Shah NS, St-Onge MP, Thacker EL, Virani SS, Voeks JH, Wang NY, Wong ND, Wong SS, Yaffe K, Martin SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2023 Update: A Report From the American Heart Association. Circulation. 2023 Feb 21;147(8):e93-e621. doi: 10.1161/CIR.0000000000001123. Epub 2023 Jan 25. PMID 36695182
- See also: World Health Organization (WHO). Noncommunicable diseases. — https://www.who.int/news-room/fact-sheets/detail/noncommunicable-diseases
- See also: Risk Factors for Coronary Artery Disease — https://www.ncbi.nlm.nih.gov/books/NBK554410/
- See also: Conselho Federal de Enfermagem - COFEN. Código de Ética dos Profissionais de Enfermagem. — https://www.cofen.gov.br/resolucao-cofen-no-5642017/
- See also: World Health Organization (WHO). Global strategy on digital health 2020-2025. — https://www.who.int/docs/default-source/documents/gs4dhdaa2a9f352b0445bafbc79ca799dce4d.pdf
- See also: Brasil. Ministério da Saúde (MS). Estratégia de Saúde Digital para o Brasil 2020-2028. — https://bvsms.saude.gov.br/bvs/publicacoes/estrategia_saude_digital_Brasil.pdf
- See also: Brasil. Lei n° 14.510, de 27 de dezembro de 2022. Altera a Lei nº 8.080, de 19 de setembro de 1990, para autorizar e disciplinar a prática da telessaúde em todo o território nacional. — https://legis.senado.leg.br/norma/36665930/publicacao/36672979
- See also: Brasil. Portaria GM/MS n° 635, de 22 de maio de 2023. Institui, define e cria incentivo financeiro federal de implantação, custeio e desempenho para as modalidades de equipes Multiprofissionais na Atenção Primária à Saúde. — https://www.in.gov.br/en/web/dou/-/portaria-gm/ms-n-635-de-22-de-maio-de-2023-484773799
- See also: Organização Pan-Americana de Saúde (OPAS). Organização Mundial da Saúde. Teleconsulta durante uma pandemia. — https://www.paho.org/ish/images/docs/covid-19-teleconsultas-pt.pdf?ua=1
- See also: Conselho Federal de Enfermagem (COFEN). Resolução n° 634/2020. Autoriza e normatiza a teleconsulta de enfermagem como forma de combate à pandemia provocada pelo novo coronavírus (Sars-Cov-2) — https://www.cofen.gov.br/resolucao-cofen-no-0634-2020/
- See also: Conselho Federal de Enfermagem (COFEN). Resolução n° 696/2022. Dispõe sobre a atuação da Enfermagem na Saúde Digital, normatizando a Telenfermagem. — https://www.cofen.gov.br/wp-content/uploads/2022/05/Resolucao-696-2022.pdf
- See also: Conselho Federal de Enfermagem (COFEN). Resolução COFEN nº 736/2024. Dispõe sobre a implementação do Processo de Enfermagem em todo contexto socioambiental onde ocorre o cuidado de enfermagem. — https://www.cofen.gov.br/resolucao-cofen-no-736-de-17-de-janeiro-de-2024/
- See also: National Institute for Health Research (NIHR). Patient and public involvement in health and social care research: a handbook for researchers. — https://oxfordbrc.nihr.ac.uk/wp-content/uploads/2017/03/RDS-PPI-Handbook-2014-v8-FINAL-2.pdf
- See also: Ebook - Envolvimento do paciente e do público em pesquisas — https://repositorio.ufrn.br/handle/123456789/59058
- See also: Conselho Nacional de Saúde (BR). Resolução nº 466, de 12 de dezembro de 2012. — https://conselho.saude.gov.br/resolucoes/2012/Reso466.pdf